CLINICAL TRIAL: NCT03201406
Title: Retrospective Analysis of Renal Prognosis in Patients With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201612068RIND
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Diabetic Nephropathies; Lupus Nephritis; Rapidly Progressive Glomerulonephritis; Chronic Kidney Diseases
Keywords: Renal biopsy, Chronic kidney disease,Diabetic nephropathy,Lupus Nephritis
MeSH Terms: conditions — Diabetic Nephropathies; Lupus Nephritis; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
During 1993 and 2006, a total of 987 patients older than 20 years underwent native kidney biopsy at the Renal Division of this hospital. 404 patients with membranoproliferative glomerulonephritis and mesangioproliferative glomerulonephritis, and patients with secondary glomerulonephritis or other renal pathologies, such as diabetic nephropathy, lupus nephritis, rapid progress glomerulonephritis, acute tubular necrosis, and tubulointerstitial nephritis will be analyzed. The demographic characteristics and laboratory data of these patients at presentation or before renal biopsy will be recorded. These data included parameters such as age, sex, diabetes, hypertension, immunosuppressants treatment, BUN, serum creatinine, albumin, hemoglobin, total cholesterol, triglycerides, and urine protein. All subjects will be followed until 2015 for occurrence of primary endpoints, including all-cause death or ESRD requiring long-term dialysis or renal transplantation. A total of 433 patients who had been followed for 3 years during 2003 and 2007 will receive regular clinic follow-up. GFR will be estimated according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula: 186 x Scr -1.154 x age -0.203 x 0.742 (if female). CKD stage will be determined as described by the National Kidney Foundation of the United States. At the time of entry, GFRs of 30-59, 29-15 and < 15 ml/min/1.73 m2 for more than 3 months will be classified as CKD stages 3, 4 and 5, respectively. Baseline Data of the 433 patients are used as recorded at the beginning during 2003 and 2007. The observation period of each patient is defined to start immediately after the registered measurement of serum creatinine satisfying the above criteria (designated as the index date) and lasted until ESRD or end of 2015. ESRD is defined as initiation of RRT, i.e. chronic dialysis or renal transplantation.

ELIGIBILITY:
Inclusion Criteria :

* Patients older than 20 years.
* Patients underwent native kidney biopsy at the Renal Division of this hospital, and with renal pathologies, such as diabetic nephropathy, lupus nephritis, rapid progress glomerulonephritis.
* Patients were classified as CKD stages 3A, 3B, 4 and 5 at the time of entry.

Exclusion Criteria :

* Patients younger than 20 years.
* Patients older than 20 years underwent native kidney biopsy at the Renal Division of this hospital, and with renal pathologies, such as membranoproliferative glomerulonephritis, mesangioproliferative glomerulonephritis, secondary glomerulonephritis, or other renal pathologies, such as, acute tubular necrosis, and tubulointerstitial nephritis.
* Patients older than 20 years but eGFR ≧ 60 ml/min/1.73 m2 at the time of entry.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Center cases
Sampling Method: Non-Probability Sample
Enrollment: 837 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
End Stage Renal Disease | 21 years
Mortality | 21 years

CONTACTS AND LOCATIONS:
Overall Officials: YUNG-MING CHEN, M.D., Principal Investigator — Attending Physician, Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan, ROC
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Yung-Ming Chen, Taipei